CLINICAL TRIAL: NCT05855915
Title: Effectiveness of Kinesio Taping Versus Sham Taping Along With Routine Physical Therapy Among Patients of Chronic Low Back Pain A Randomised Trial
Brief Title: Effectiveness of KT VS ST Along With Routine Physical Therapy Among Patients of Chronic Low Back Pain RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DPT/Batch-Fall18/523
Record Dates: First submitted 2023-03-15; First posted 2023-05-12 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesio taping (Experimental): Kinesotaping will be applied with routine physical therapy
  Interventions: Diagnostic Test: Kinesio taping
- Sham taping (Experimental): Sham taping will be applied with routine physical therapy
  Interventions: Diagnostic Test: Sham taping

INTERVENTIONS:
Diagnostic Test: Kinesio taping — Kinesotaping will be applied with routine physical therapy
  Arms: Kinesio taping
Diagnostic Test: Sham taping — Sham taping will be applied with routine physical therapy
  Arms: Sham taping

SUMMARY:
To determine the effectiveness of Kineso taping (KT) Versus Sham taping along with routine physical therapy among Chronic Low Back pain (CLBP) patients.

ELIGIBILITY:
Inclusion Criteria:

Pain in the area between 12 ribs and hip crease with or without leg pain. Age ranges from 18 to 65 years. Low back pain for 6 weeks. Moderate pain intensity with pain score.

Exclusion Criteria:

Known or suspected Spinal lesions. Spinal surgery within first 6 months. Physical Therapy for low back pain for past 6 months. Severe Complications.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Oswestry Disability Index | 6 Months

CONTACTS AND LOCATIONS:
Locations (1):
- Chaudary Muhammad Akram Teaching Hospital, Azra Naheed Medical College, Superior University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No